CLINICAL TRIAL: NCT00604786
Title: Pilot Study of the Effect of Omalizumab on Basophil and Mast Responses to Intranasal Cat Allergen Challenge
Brief Title: The Effect of Omalizumab on Responses to Cat Allergen Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00007520; U19AI070345 (NIH)
Record Dates: First submitted 2008-01-04; First posted 2008-01-30 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Allergic Rhinitis
Keywords: Basophils; Mast Cells; IgE; IgE receptors; omalizumab
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omalizumab subcutaneous (Experimental): This active are will receive treatment with omalizumab subcutaneously at the dose currently FDA-approved for the treatment of allergic asthma. There is a weight and IgE based dosing table in the and subjects receive therapy by subcutaneous injection every 2 or 4 weeks. The lower range of dosing is 150 mg q 4weeks ( one injection) with the upper range 375 mg every 2 weeks ( three injections).
  The dosing is based on IgE levels and IGE and is given by subcutaneous injection every 2 to 4 weeks
  Interventions: Drug: omalizumab
- Placebo Subcutaneous (Placebo Comparator): This placebo arm will receive identical treatment with placebo injections subcutaneously at the dose currently FDA-approved for the treatment of allergic asthma. There is a weight and IgE based dosing table in the and subjects receive therapy by subcutaneous injection every 2 or 4 weeks. The lower range of dosing is 150 mg q 4weeks ( one injection) with the upper range 375 mg every 2 weeks ( three injections).
  The dosing is based on IgE levels and IGE and is given by subcutaneous injection every 2 to 4 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omalizumab — Dosing is based on IgE level and weight given every 2 or 4 weeks
  Other Names: Xolair
  Arms: Omalizumab subcutaneous
Drug: placebo — Dosing is based on IgE level and weight given every 2 or 4 weeks
  Arms: Placebo Subcutaneous

SUMMARY:
This research is being done to study the effects of the drug omalizumab (Xolair) in people with cat allergies. The investigators will use omalizumab to study changes in the cells in the nose, skin and blood that cause allergies. The investigators predict that cells in the blood will be effected before cells in the nose or skin.

DETAILED DESCRIPTION:
Omalizumab is a monoclonal antibody directed against Immunoglobulin E (IgE) and is FDA-approved for use in allergic asthma, though its clinical role is not precisely defined. It binds IgE on the same site of the Fc domain as the high affinity IgE receptor (FcεRI), and therefore, blocks the interaction between IgE and mast cells or basophils. It, therefore, may be used as a mechanistic tool in the study of IgE. As IgE levels are reduced with omalizumab, FcεRI expression on human basophils is reduced. This reduction of basophil receptors and allergen induced activation is pronounced within 7 days of the initial administration and is reversible once omalizumab administration is discontinued. The omalizumab-induced reductions in mast cell FcεRI expression and function is unchanged at day 7 and significantly reduced by day 70. These changes were based upon intravenously administered omalizumab at a dose of 0.03 mg/kg/IU IgE/mL in a total of three subjects. We propose to exploit the kinetics of faster omalizumab effects on circulating basophils relative to tissue mast cells to elucidate the role of the basophil versus mast cell activation in nasal airway allergen challenge, which has not been studied to date.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide informed consent
* Male or Female (non-pregnant), age 18-50
* Females must be: Surgically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation), OR postmenopausal (at least 1 year since last menses), OR using a medically acceptable form of birth control throughout the duration of the study.
* Clinical history of seasonal or perennial allergic rhinitis for at least two years, with or without mild persistent asthma
* Positive puncture skin test greater than or equal to 5 mm diluent control
* Positive Immunocap to Fel d 1 > 0.35 kallikrein unit/L
* Positive intranasal cat allergen challenge as defined by > 5 sneezes or a tripling of measured nasal lavage mediators
* In vitro assay of basophil responsiveness to cat allergen with greater than 20% histamine release
* The use of antihistamines, cromolyn, leukotriene modifiers and other non-steroid (astelin and topical decongestants), nasal medications will be allowed, but they will be withheld for 5 days prior to each nasal allergen provocation session. Inhaled corticosteroids for mild asthma will be permissible.
* No known contraindications to therapy with omalizumab

Exclusion Criteria:

* Asthma with forced expiratory volume at one second (FEV1) < 80%, moderate to severe asthma classification per National Asthma Education and Prevention Program Expert Panel (NAEP) Standards (1997 National Asthma Education and Prevention Program Expert Panel Report II guidelines)
* Serum IgE levels less than 30 IU/mL or greater than 700 IU/mL at the time of enrollment will be excluded
* Unexplained elevation of erythrocyte sedimentation rate (ESR), hematocrit < 32%, white blood cell (WBC) count 2400/microliter lower limit of normal, platelet < 75000/microliter, creatinine > 141.4 micromolar/L, or aspartate aminotransferase (AST) > 100 IU/L
* Body weight less than 30 kg or greater than 150 kg will be excluded.
* Plans to become pregnant or breastfeed will be excluded from the study
* A perforated nasal septum, structural nasal defect, large nasal polyps causing obstruction, evidence of acute or chronic sinusitis
* A life expectancy less than 6 months
* A terminal illness as determined by the investigator
* A history of malignancy, anaphylaxis or bleeding disorder are also exclusion illnesses.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Use of any investigational drugs within 8 weeks of participation
* Contraindications to omalizumab include patients with a previous hypersensitivity to omalizumab
* Recent recipient of any licensed or investigational live attenuated vaccine(s) within two months of study initiation such as flu mist.
* Prior use of omalizumab
* Frequent sinusitis (>2/ documented episodes per year) or active sinusitis within 2 weeks of enrollment
* Use of immunotherapy within the last 5 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarbjit S Saini, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Strunk RC, Bloomberg GR. Omalizumab for asthma. N Engl J Med. 2006 Jun 22;354(25):2689-95. doi: 10.1056/NEJMct055184. No abstract available. PMID 16790701
- [Background] Presta LG, Lahr SJ, Shields RL, Porter JP, Gorman CM, Fendly BM, Jardieu PM. Humanization of an antibody directed against IgE. J Immunol. 1993 Sep 1;151(5):2623-32. PMID 8360482
- [Background] Schulman ES. Development of a monoclonal anti-immunoglobulin E antibody (omalizumab) for the treatment of allergic respiratory disorders. Am J Respir Crit Care Med. 2001 Oct 15;164(8 Pt 2):S6-11. doi: 10.1164/ajrccm.164.supplement_1.2103025. PMID 11704611
- [Background] MacGlashan DW Jr, Bochner BS, Adelman DC, Jardieu PM, Togias A, McKenzie-White J, Sterbinsky SA, Hamilton RG, Lichtenstein LM. Down-regulation of Fc(epsilon)RI expression on human basophils during in vivo treatment of atopic patients with anti-IgE antibody. J Immunol. 1997 Feb 1;158(3):1438-45. PMID 9013989
- [Background] Saini SS, MacGlashan DW Jr, Sterbinsky SA, Togias A, Adelman DC, Lichtenstein LM, Bochner BS. Down-regulation of human basophil IgE and FC epsilon RI alpha surface densities and mediator release by anti-IgE-infusions is reversible in vitro and in vivo. J Immunol. 1999 May 1;162(9):5624-30. PMID 10228046
- [Background] Beck LA, Marcotte GV, MacGlashan D, Togias A, Saini S. Omalizumab-induced reductions in mast cell Fce psilon RI expression and function. J Allergy Clin Immunol. 2004 Sep;114(3):527-30. doi: 10.1016/j.jaci.2004.06.032. PMID 15356552
- [Background] Proud D, Bailey GS, Naclerio RM, Reynolds CJ, Cruz AA, Eggleston PA, Lichtenstein LM, Togias AG. Tryptase and histamine as markers to evaluate mast cell activation during the responses to nasal challenge with allergen, cold, dry air, and hyperosmolar solutions. J Allergy Clin Immunol. 1992 Jun;89(6):1098-110. doi: 10.1016/0091-6749(92)90293-b. PMID 1607547
- [Background] Nathan RA, Eccles R, Howarth PH, Steinsvag SK, Togias A. Objective monitoring of nasal patency and nasal physiology in rhinitis. J Allergy Clin Immunol. 2005 Mar;115(3 Suppl 1):S442-59. doi: 10.1016/j.jaci.2004.12.015. PMID 15746882
- [Background] Naclerio RM, Proud D, Togias AG, Adkinson NF Jr, Meyers DA, Kagey-Sobotka A, Plaut M, Norman PS, Lichtenstein LM. Inflammatory mediators in late antigen-induced rhinitis. N Engl J Med. 1985 Jul 11;313(2):65-70. doi: 10.1056/NEJM198507113130201. PMID 2582257
- [Background] Lin H, Boesel KM, Griffith DT, Prussin C, Foster B, Romero FA, Townley R, Casale TB. Omalizumab rapidly decreases nasal allergic response and FcepsilonRI on basophils. J Allergy Clin Immunol. 2004 Feb;113(2):297-302. doi: 10.1016/j.jaci.2003.11.044. PMID 14767445
- [Background] Hanf G, Noga O, O'Connor A, Kunkel G. Omalizumab inhibits allergen challenge-induced nasal response. Eur Respir J. 2004 Mar;23(3):414-8. doi: 10.1183/09031936.04.00024504. PMID 15065831
- [Background] Corren J, Diaz-Sanchez D, Saxon A, Deniz Y, Reimann J, Sinclair D, Davancaze T, Adelman D. Effects of omalizumab, a humanized monoclonal anti-IgE antibody, on nasal reactivity to allergen and local IgE synthesis. Ann Allergy Asthma Immunol. 2004 Sep;93(3):243-8. doi: 10.1016/S1081-1206(10)61495-0. PMID 15478383
- [Background] Pods R, Ross D, van Hulst S, Rudack C, Maune S. RANTES, eotaxin and eotaxin-2 expression and production in patients with aspirin triad. Allergy. 2003 Nov;58(11):1165-70. doi: 10.1034/j.1398-9995.2003.00276.x. PMID 14616128
- [Background] Berkman N, Ohnona S, Chung FK, Breuer R. Eotaxin-3 but not eotaxin gene expression is upregulated in asthmatics 24 hours after allergen challenge. Am J Respir Cell Mol Biol. 2001 Jun;24(6):682-7. doi: 10.1165/ajrcmb.24.6.4301. PMID 11415932
- [Background] Salib RJ, Lau LC, Howarth PH. Nasal lavage fluid concentrations of eotaxin-1 (CCL11) in naturally occurring allergic rhinitis: relationship to disease activity, nasal luminal eosinophil influx, and plasma protein exudation. Clin Exp Allergy. 2005 Aug;35(8):995-1002. doi: 10.1111/j.1365-2222.2005.02236.x. PMID 16120080
- [Background] Terada N, Hamano N, Kim WJ, Hirai K, Nakajima T, Yamada H, Kawasaki H, Yamashita T, Kishi H, Nomura T, Numata T, Yoshie O, Konno A. The kinetics of allergen-induced eotaxin level in nasal lavage fluid: its key role in eosinophil recruitment in nasal mucosa. Am J Respir Crit Care Med. 2001 Aug 15;164(4):575-9. doi: 10.1164/ajrccm.164.4.2009046. PMID 11520718
- [Background] Ong YE, Menzies-Gow A, Barkans J, Benyahia F, Ou TT, Ying S, Kay AB. Anti-IgE (omalizumab) inhibits late-phase reactions and inflammatory cells after repeat skin allergen challenge. J Allergy Clin Immunol. 2005 Sep;116(3):558-64. doi: 10.1016/j.jaci.2005.05.035. PMID 16159624
- [Background] Bousquet J, Cabrera P, Berkman N, Buhl R, Holgate S, Wenzel S, Fox H, Hedgecock S, Blogg M, Cioppa GD. The effect of treatment with omalizumab, an anti-IgE antibody, on asthma exacerbations and emergency medical visits in patients with severe persistent asthma. Allergy. 2005 Mar;60(3):302-8. doi: 10.1111/j.1398-9995.2004.00770.x. PMID 15679714
- [Background] Humbert M, Beasley R, Ayres J, Slavin R, Hebert J, Bousquet J, Beeh KM, Ramos S, Canonica GW, Hedgecock S, Fox H, Blogg M, Surrey K. Benefits of omalizumab as add-on therapy in patients with severe persistent asthma who are inadequately controlled despite best available therapy (GINA 2002 step 4 treatment): INNOVATE. Allergy. 2005 Mar;60(3):309-16. doi: 10.1111/j.1398-9995.2004.00772.x. PMID 15679715
- [Background] Casale TB. Anti-immunoglobulin E (omalizumab) therapy in seasonal allergic rhinitis. Am J Respir Crit Care Med. 2001 Oct 15;164(8 Pt 2):S18-21. doi: 10.1164/ajrccm.164.supplement_1.2103023. PMID 11704613
- [Background] Adelroth E, Rak S, Haahtela T, Aasand G, Rosenhall L, Zetterstrom O, Byrne A, Champain K, Thirlwell J, Cioppa GD, Sandstrom T. Recombinant humanized mAb-E25, an anti-IgE mAb, in birch pollen-induced seasonal allergic rhinitis. J Allergy Clin Immunol. 2000 Aug;106(2):253-9. doi: 10.1067/mai.2000.108310. PMID 10932067
- [Background] Chervinsky P, Casale T, Townley R, Tripathy I, Hedgecock S, Fowler-Taylor A, Shen H, Fox H. Omalizumab, an anti-IgE antibody, in the treatment of adults and adolescents with perennial allergic rhinitis. Ann Allergy Asthma Immunol. 2003 Aug;91(2):160-7. doi: 10.1016/S1081-1206(10)62171-0. PMID 12952110
- [Background] Kuehr J, Brauburger J, Zielen S, Schauer U, Kamin W, Von Berg A, Leupold W, Bergmann KC, Rolinck-Werninghaus C, Grave M, Hultsch T, Wahn U. Efficacy of combination treatment with anti-IgE plus specific immunotherapy in polysensitized children and adolescents with seasonal allergic rhinitis. J Allergy Clin Immunol. 2002 Feb;109(2):274-80. doi: 10.1067/mai.2002.121949. PMID 11842297
- [Background] Casale TB, Bernstein IL, Busse WW, LaForce CF, Tinkelman DG, Stoltz RR, Dockhorn RJ, Reimann J, Su JQ, Fick RB Jr, Adelman DC. Use of an anti-IgE humanized monoclonal antibody in ragweed-induced allergic rhinitis. J Allergy Clin Immunol. 1997 Jul;100(1):110-21. doi: 10.1016/s0091-6749(97)70202-1. PMID 9257795
- [Background] Deniz YM, Gupta N. Safety and tolerability of omalizumab (Xolair), a recombinant humanized monoclonal anti-IgE antibody. Clin Rev Allergy Immunol. 2005 Aug;29(1):31-48. doi: 10.1385/criai:29:1:031. PMID 16222082
- [Derived] Paterniti M, Kelly DC, Eckman JA, Sterba PM, Hamilton RG, Bochner BS, Macglashan DW Jr, Saini SS. Cat allergen-induced blood basophil reactivity in vitro predicts acute human nasal allergen challenge responses in vivo. Clin Exp Allergy. 2011 Jul;41(7):963-9. doi: 10.1111/j.1365-2222.2011.03719.x. Epub 2011 Mar 29. PMID 21668817

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab Subcutaneous: This active are will receive treatment with omalizumab subcutaneously at the dose currently FDA-approved for the treatment of allergic asthma. There is a weight and immunoglobulin E (IgE) based dosing table in the and subjects receive therapy by subcutaneous injection every 2 or 4 weeks. The lower range of dosing is 150 mg q 4weeks ( one injection) with the upper range 375 mg every 2 weeks ( three injections).
  The dosing is based on IgE levels and IGE and is given by subcutaneous injection every 2 to 4 weeks
Period: Overall Study
Arm/Group | Omalizumab Subcutaneous | Placebo Subcutaneous
Started | 14 | 4
Completed | 12 | 4
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: This arm will receive treatment with omalizumab at the dose FDA-approved for the treatment of allergic asthma.
  omalizumab: IgE 30-100 int. units/mL: 30-90 kg: 150 mg every 4 weeks >90-150 kg: 300 mg every 4 weeks
  IgE >100-200 int. units/mL:
  30-90 kg: 300 mg every 4 weeks >90-150 kg: 225 mg every 2 weeks
  IgE >200-300 int. units/mL:
  30-60 kg: 300 mg every 4 weeks >60-90 kg: 225 mg every 2 weeks >90-150 kg: 300 mg every 2 weeks
  IgE >300-400 int. units/mL:
  30-70 kg: 225 mg every 2 weeks >70-90 kg: 300 mg every 2 weeks >90 kg: Do not administer dose
  IgE >400-500 int. units/mL:
  30-70 kg: 300 mg every 2 weeks >70-90 kg: 375 mg every 2 weeks >90 kg: Do not administer dose
  IgE >500-600 int. units/mL:
  30-60 kg: 300 mg every 2 weeks >60-70 kg: 375 mg every 2 weeks >70 kg: Do not administer dose
  IgE >600-700 int. units/mL:
  30-60 kg: 375 mg every 2 weeks >60 kg: Do not administer dose
- Placebo: placebo: IgE 30-100 int. units/mL: 30-90 kg: placebo every 4 weeks >90-150 kg: placebo every 4 weeks
  IgE >100-200 int. units/mL:
  30-90 kg: placebo every 4 weeks >90-150 kg: placebo every 2 weeks
  IgE >200-300 int. units/mL:
  30-60 kg: placebo every 4 weeks >60-90 kg: placebo every 2 weeks >90-150 kg: placebo every 2 weeks
  IgE >300-400 int. units/mL:
  30-70 kg: placebo every 2 weeks >70-90 kg: placebo every 2 weeks >90 kg: Do not administer dose
  IgE >400-500 int. units/mL:
  30-70 kg: placebo every 2 weeks >70-90 kg: placebo every 2 weeks >90 kg: Do not administer dose
  IgE >500-600 int. units/mL:
  30-60 kg: placebo every 2 weeks >60-70 kg: placebo every 2 weeks >70 kg: Do not administer dose
  IgE >600-700 int. units/mL:
  30-60 kg: placebo every 2 weeks >60 kg: Do not administer dose
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 14 | 4 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 4 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.6 [24 to 47] | 32.3 [25 to 49] | 31 [24 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 14 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Basophil Surface IgE
Description: Flow cytometry in mean fluorescence units.
  100%*[(3.5 month value minus baseline value)/baseline value]
Time Frame: Change from baseline to 3.5 months
Population: 2 participants on the Omalizumab subcutaneous group moved and were therefore lost to follow-up.
Measure: Mean (Standard Deviation); unit: percentage of basophil surface IgE
Arm/Group | Omalizumab Subcutaneous | Placebo Subcutaneous
Number analyzed (Participants) | 12 | 4
percentage of basophil surface IgE | -95 (3) | -10 (4)

ADVERSE EVENTS:
Time Frame: 3.5 months
Arm/Group | Omalizumab Subcutaneous | Placebo Subcutaneous
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/4
Other Adverse Events (participants affected / at risk) | 2/14 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab Subcutaneous (N=14) | Placebo Subcutaneous (N=4)
Injection site swelling (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
2 subject in active group did not finish the study, small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No